CLINICAL TRIAL: NCT05115539
Title: Assessment of Volume Status by Doppler Ultrasound to Predict Acute Kidney Injury in Critically Ill Patients
Brief Title: Assessment of Volume Status by Doppler US
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Zein Elabedeen Ahmed Abdallah, Principal Investigator, Assiut University
Other Study IDs: AVSDTPAKI
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Fluid Assessment by Doppler us Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: doppler US of portal vein, hepatic veins, intrarenal veins — Hepatic Vein Doppler : To obtain the HV PW, a phased array transducer is used with cardiac pre-sets. ECG leads are placed to assist in the interpretation of HVD in sinus rhythm as well as atrial fibrillation. The middle hepatic vein is identified from mid-subcostal or lateral views during the end-expiratory phase of the patients respiratory cycle.
  Portal vein Doppler: From a lateral costal or subcostal window, the portal vein is identified in the coronal plane using a phased-array transducer. The PV were considered abnormal if the pulsatilty index was greater than 30%. The portal pulsatility index was defined as: (VMax - VMin/VMax) * 100%. Here, VMax is the maximal velocity and VMin is the minimal velocity during the cardiac cycle.
  Intra-renal venous Doppler: From lateral costal window, the kidney is located in the coronal plane and a color flow box placed over the distal renal calyceal junction to cortex.

SUMMARY:
Fluid are used to increase cardiac output (CO) and blood pressure in patients admitted to the intensive care unit (ICU) .Fluid is an important line of therapy that needed in shocked patient, hypovolemic and following surgery to correct the volume state and avoid acute kidney injury. However, excess fluid administration may be harmful leading itself to increase rates of acute kidney injury (AKI), prolonged days of mechanical ventilation and death . Excess fluid administration may increase right and left atrial pressure leading to congestion and edema.

DETAILED DESCRIPTION:
Increasing cardiac output more than 15% following fluid administration was used as fluid responsiveness method by the Surviving Sepsis Campaign (SSC) guidelines. However, these strategies may promote over-resuscitation as most recommend continuing fluid administration until the patients are no longer VR. VR-based strategies do not assess elevations in right atrial pressure (RAP) or assess for venous congestion which could occur earlier.

The elevations of left atrial pressure can be seen clinically with hypoxia, cephalization on chest X-ray and B-lines on ultrasound resulting from pulmonary edema, while the elevation in right-sided pressure is much more difficult to detect.

It is possible that rightsided venous flow changes detect clinically important elevations in right atrial pressure that lead to venous congestion and end organ injury . Doppler flow patterns of hepatic veins (HV), portal vein (PV) and intra-renal veins (RV) are noninvasive and accurately identify early stages of right-sided venous congestion in patients who have cardiac dysfunction and congestive heart failure with elevated right atrial pressures . If HV, PV and RV can be validated as reliable measures of elevated RAP, such indicators might have utility in modulating fluid resuscitation in other critically ill patient populations.

ELIGIBILITY:
Inclusion Criteria:

* - Adult patients who admitted to critical care unit and intermediate critical care unit of Internal medicine department after obtaining consent.

Exclusion Criteria:

* 1- Children below 18 yr. 2- Patients could not be scanned within 24-h after ICU admission. 3- Patients with transplanted kidney or liver. 4- Patients with end stage renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patients who admitted to critical care unit and intermediate critical care unit of Internal medicine department after obtaining consent
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Doppler flow patterns of hepatic veins (HV), portal vein (PV) and intra-renal veins (RV) in critically ill patients and their relations to the patients' volume state. | 1 year
  hepatic veins (HV), portal vein (PV) and intra-renal veins doppler changes in critically ill patients

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Spiegel R, Teeter W, Sullivan S, Tupchong K, Mohammed N, Sutherland M, Leibner E, Rola P, Galvagno SM Jr, Murthi SB. The use of venous Doppler to predict adverse kidney events in a general ICU cohort. Crit Care. 2020 Oct 19;24(1):615. doi: 10.1186/s13054-020-03330-6. PMID 33076961